CLINICAL TRIAL: NCT01758354
Title: Newborn Screening Assay of Pompe's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 9461700818
Record Dates: First submitted 2008-07-09; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-11

CONDITIONS: Pompe Disease
Keywords: Pompe disease; alpha glucosidase deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pompe disease newborn screening (Experimental): newborns will be tested if they were affected by Pompe disease
  Interventions: Other: Pompe disease newborn screening

INTERVENTIONS:
Other: Pompe disease newborn screening — DBS will be tested for acid alpha-glucosidase (GAA)activity. Newborns with low GAA activity will received a confirmatory blood sampling and clinical evaluation for the presence of cardiomyopathy.

SUMMARY:
The purpose of this study is to test the feasibility of a newborn screen assay for Pompe disease

DETAILED DESCRIPTION:
DBS from newborn will be tested for acid alpha-glucosidase (GAA) activity. Babies with low GAA activity will be confirmed for Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* newborns receiving newborn screening in Newborn Screening center of National Taiwan Univeristy Hospital
* parents signed inform consent for this study

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 236536 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
detect patients with infantile onset Pompe disease | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Whu-Liang Hwu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan